CLINICAL TRIAL: NCT03343886
Title: Ageing and Health. Spanish Longitudinal Study on Ageing, Physical and Mental Health, and Its Determinants
Brief Title: Ageing and Health. Spanish Longitudinal Study
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Fundació Sant Joan de Déu (Other); Universidad Autonoma de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: COURAGE2020; FP7/2007-2013- 316795 (Other Grant/Funding Number: European Commission); ACI2009-1010 (Other Grant/Funding Number: Spanish Ministry of Science and Innovation); PS09/00295 (Other Grant/Funding Number: Carlos III Health Institute); PS09/01845 (Other Grant/Funding Number: Carlos III Health Institute); PI12/01490 (Other Grant/Funding Number: Carlos III Health Institute); PI13/00059 (Other Grant/Funding Number: Carlos III Health Institute); PI16/01073 (Other Grant/Funding Number: Carlos III Health Institute); PI16/00812 (Other Grant/Funding Number: Carlos III Health Institute); PI19/00088 (Other Grant/Funding Number: Carlos III Health Institute); PI19/00103 (Other Grant/Funding Number: Carlos III Health Institute); PI19/00150 (Other Grant/Funding Number: Carlos III Health Institute); PI19/00235 (Other Grant/Funding Number: Carlos III Health Institute); PI22/00309 (Other Grant/Funding Number: Carlos III Health Institute); PI22/00340 (Other Grant/Funding Number: Carlos III Health Institute); PI22/00374 (Other Grant/Funding Number: Carlos III Health Institute); PI22/00375 (Other Grant/Funding Number: Carlos III Health Institute)
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Health, Subjective; Disability, Evaluation; Chronic Disease; Mental Disorder; Aging; Loneliness; Well-being; Cognitive Decline
Keywords: Health Status; Well-being; Mental Health; Risk Factors; Aging
MeSH Terms: conditions — Chronic Disease; Mental Disorders; Cognitive Dysfunction; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 2011: A nationally representative sample of 4753 non-institutionalized adults aged 18 years or older from the Spanish population was collected (with an over-sampling of people aged 50+ years). A multi-stage clustered design was employed. A total of 2528 individuals were re-interviewed in 2014. In 2018, 1577 were again evaluated. Finally, in 2022, 963 participants took part of another study's evaluation.
- Cohort 2019: 3002 participants from the regions of Madrid and Barcelona were brought in between 2019 and 2021. They are now under a second evaluation (2023). In 2020, during the first Coronavirus (COVID-19) lockdown, 1166 of the participants from the first wave of the cohort was telephonically interviewed, a lateral sub-study evaluation.

SUMMARY:
Age with Health is a longitudinal cohort study aimed to examine trajectories of health, disability and wellbeing and their determinants for Spanish ageing population. The data that makes up the baseline was collected from a nationally representative sample of non-institutionalized adults as part of the "Collaborative Research on Aging in Europe (COURAGE in Europe)" project between July 2011 and May 2012. The second wave was carried out as part of the "Age with Health" project between December 2014 and June 2015, and three years later, in 2018, the third wave was carried out. In 2019-2021, a new cohort of participants were brought in (2019 cohort), some of whom were interviewed again by telephone during the first Coronavirus (COVID-19) lockdown, in early 2020. During 2022 a new evaluation of the participants of both cohorts (2011 and 2019) is expected.

DETAILED DESCRIPTION:
Study Design:

A prospective cohort general population study.

Sample:

Wave 1: A nationally representative sample of non-institutionalized adults aged 18 years or older from the Spanish population was collected (with an over-sampling of people aged 50+ years). A multi-stage clustered design was employed; four strata based on the number of inhabitants of the municipalities were built for each of the 17 Spanish autonomous communities. Clusters were selected within the strata with a probability of inclusion relative to their size. Within each cluster, households were randomly selected from a list of all households. In case there was more than one individual from the corresponding age group in the household, a random method was employed to select the individual participant.

Wave 2: Wave 1 sample was re-interviewed (Wave 2) in 2014-2015.

Wave 3: in 2018, participants were again evaluated. Complementarily, between 2019 and 2021 a new sample from the regions of Madrid and Barcelona were brought in, and it was interviewed again by telephone during the first COVID-19 lockdown, in May-June 2020.

Wave 4: a new evaluation of the participants of both cohorts 2011 and 2019 was carried out, in the fist case it terminated in 2022, while the data collection for 2019 cohort is still going on, expected to terminate for December 2023.

Wave 5: a new and last evaluation is expected for both cohort in 2025.

Data collection:

Face-to-face interviews by Computer-Assisted Personal Interviewing at the respondents' homes by trained interviewers. All interviewers received a standardized training. Data quality control was also performed. A proxy interview was administered in those cases in which the participant presents physical or cognitive limitations that may impede the correct administration of the individual interview.

Main project objectives:

To assess trajectories of general health, disability and well-being in Spanish ageing population.

Secondary objectives:

To identify trajectories of healthy ageing (in terms of physical health, mental health, functioning and well-being) in Spanish adult population as well as their determinants To analyse prevalence and impact of chronic health conditions, mental health problems, well-being and loneliness on mortality in Spanish adult population.

To determine risk factors for incidence and persistence of mental and physical health problems in Spanish ageing population.

Main project hypotheses:

The trajectories of health, functioning and well-being will be encompassed by relevant environmental factors such as social support, loneliness and health care utilization, personal factors (socio-demographic characteristics, healthy lifestyles, and high cognitive reserve among others) and other biological and health-related factors (weight, height, waist circumference, executive functions, blood pressure, grip strength, vision acuity, presence of mental and physical health problems and quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized Spanish residents
* 18 years and over

Exclusion Criteria:

* Institutionalized population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-living individuals in Spain aged 18 years or older
Sampling Method: Probability Sample
Enrollment: 7755 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Ayuso Mateos, MD, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (3):
- Spain (3):
  - Fundació Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - Fundación de Investigación Biomédica - Hospital Universitario de La Princesa, Madrid
  - Universidad Autónoma de Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Undecided
A sharing plan description has to be still agreed between the different Principal Investigators

REFERENCES:
- [Result] Miret M, Caballero FF, Olaya B, Koskinen S, Naidoo N, Tobiasz-Adamczyk B, Leonardi M, Haro JM, Chatterji S, Ayuso-Mateos JL. Association of experienced and evaluative well-being with health in nine countries with different income levels: a cross-sectional study. Global Health. 2017 Aug 23;13(1):65. doi: 10.1186/s12992-017-0290-0. PMID 28835255
- [Result] Olaya B, Moneta MV, Domenech-Abella J, Miret M, Bayes I, Ayuso-Mateos JL, Haro JM. Mobility Difficulties, Physical Activity, and All-cause Mortality Risk in a Nationally representative Sample of Older Adults. J Gerontol A Biol Sci Med Sci. 2018 Aug 10;73(9):1272-1279. doi: 10.1093/gerona/glx121. PMID 28633439
- [Result] Lara E, Koyanagi A, Domenech-Abella J, Miret M, Ayuso-Mateos JL, Haro JM. The Impact of Depression on the Development of Mild Cognitive Impairment over 3 Years of Follow-Up: A Population-Based Study. Dement Geriatr Cogn Disord. 2017;43(3-4):155-169. doi: 10.1159/000455227. Epub 2017 Feb 9. PMID 28178703
- [Result] Martin-Maria N, Miret M, Caballero FF, Rico-Uribe LA, Steptoe A, Chatterji S, Ayuso-Mateos JL. The Impact of Subjective Well-being on Mortality: A Meta-Analysis of Longitudinal Studies in the General Population. Psychosom Med. 2017 Jun;79(5):565-575. doi: 10.1097/PSY.0000000000000444. PMID 28033196
- [Result] Lara E, Koyanagi A, Caballero F, Domenech-Abella J, Miret M, Olaya B, Rico-Uribe L, Ayuso-Mateos JL, Haro JM. Cognitive reserve is associated with quality of life: A population-based study. Exp Gerontol. 2017 Jan;87(Pt A):67-73. doi: 10.1016/j.exger.2016.10.012. Epub 2016 Nov 5. PMID 27825839
- [Result] Kamenov K, Caballero FF, Miret M, Leonardi M, Sainio P, Tobiasz-Adamczyk B, Haro JM, Chatterji S, Ayuso-Mateos JL, Cabello M. Which Are the Most Burdensome Functioning Areas in Depression? A Cross-National Study. Front Psychol. 2016 Aug 31;7:1342. doi: 10.3389/fpsyg.2016.01342. eCollection 2016. PMID 27630609
- [Result] Martin-Maria N, Caballero FF, Olaya B, Rodriguez-Artalejo F, Haro JM, Miret M, Ayuso-Mateos JL. Positive Affect Is Inversely Associated with Mortality in Individuals without Depression. Front Psychol. 2016 Jul 12;7:1040. doi: 10.3389/fpsyg.2016.01040. eCollection 2016. PMID 27462289
- [Result] Raggi A, Corso B, Minicuci N, Quintas R, Sattin D, De Torres L, Chatterji S, Frisoni GB, Haro JM, Koskinen S, Martinuzzi A, Miret M, Tobiasz-Adamczyk B, Leonardi M. Determinants of Quality of Life in Ageing Populations: Results from a Cross-Sectional Study in Finland, Poland and Spain. PLoS One. 2016 Jul 19;11(7):e0159293. doi: 10.1371/journal.pone.0159293. eCollection 2016. PMID 27434374
- [Result] Tyrovolas S, Koyanagi A, Olaya B, Ayuso-Mateos JL, Miret M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM. Factors associated with skeletal muscle mass, sarcopenia, and sarcopenic obesity in older adults: a multi-continent study. J Cachexia Sarcopenia Muscle. 2016 Jun;7(3):312-21. doi: 10.1002/jcsm.12076. Epub 2015 Oct 7. PMID 27239412
- [Result] Lara E, Koyanagi A, Olaya B, Lobo A, Miret M, Tyrovolas S, Ayuso-Mateos JL, Haro JM. Mild cognitive impairment in a Spanish representative sample: prevalence and associated factors. Int J Geriatr Psychiatry. 2016 Aug;31(8):858-67. doi: 10.1002/gps.4398. Epub 2016 Feb 28. PMID 26923809
- [Result] Olaya B, Moneta MV, Koyanagi A, Lara E, Miret M, Ayuso-Mateos JL, Chatterji S, Leonardi M, Koskinen S, Tobiasz-Adamczyk B, Lobo A, Haro JM. The joint association of depression and cognitive function with severe disability among community-dwelling older adults in Finland, Poland and Spain. Exp Gerontol. 2016 Apr;76:39-45. doi: 10.1016/j.exger.2016.01.010. Epub 2016 Jan 22. PMID 26805608
- [Result] Rico-Uribe LA, Caballero FF, Olaya B, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM, Chatterji S, Ayuso-Mateos JL, Miret M. Loneliness, Social Networks, and Health: A Cross-Sectional Study in Three Countries. PLoS One. 2016 Jan 13;11(1):e0145264. doi: 10.1371/journal.pone.0145264. eCollection 2016. PMID 26761205
- [Result] Tyrovolas S, Koyanagi A, Olaya B, Ayuso-Mateos JL, Miret M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM. The role of muscle mass and body fat on disability among older adults: A cross-national analysis. Exp Gerontol. 2015 Sep;69:27-35. doi: 10.1016/j.exger.2015.06.002. Epub 2015 Jun 3. PMID 26048566
- [Result] Koyanagi A, Stickley A, Garin N, Miret M, Ayuso-Mateos JL, Leonardi M, Koskinen S, Galas A, Haro JM. The association between obesity and back pain in nine countries: a cross-sectional study. BMC Public Health. 2015 Feb 11;15:123. doi: 10.1186/s12889-015-1362-9. PMID 25886589
- [Result] Tyrovolas S, Koyanagi A, Garin N, Olaya B, Ayuso-Mateos JL, Miret M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM. Diabetes mellitus and its association with central obesity and disability among older adults: a global perspective. Exp Gerontol. 2015 Apr;64:70-7. doi: 10.1016/j.exger.2015.02.010. Epub 2015 Feb 16. PMID 25688991
- [Result] Tyrovolas S, Koyanagi A, Garin N, Olaya B, Ayuso-Mateos JL, Miret M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM. Determinants of the components of arterial pressure among older adults--the role of anthropometric and clinical factors: a multi-continent study. Atherosclerosis. 2015 Feb;238(2):240-9. doi: 10.1016/j.atherosclerosis.2014.11.029. Epub 2014 Dec 9. PMID 25528433
- [Result] Miret M, Caballero FF, Chatterji S, Olaya B, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Haro JM, Ayuso-Mateos JL. Health and happiness: cross-sectional household surveys in Finland, Poland and Spain. Bull World Health Organ. 2014 Oct 1;92(10):716-25. doi: 10.2471/BLT.13.129254. Epub 2014 Aug 13. PMID 25378725
- [Result] Garin N, Olaya B, Moneta MV, Miret M, Lobo A, Ayuso-Mateos JL, Haro JM. Impact of multimorbidity on disability and quality of life in the Spanish older population. PLoS One. 2014 Nov 6;9(11):e111498. doi: 10.1371/journal.pone.0111498. eCollection 2014. PMID 25375890
- [Result] Garin N, Olaya B, Miret M, Ayuso-Mateos JL, Power M, Bucciarelli P, Haro JM. Built environment and elderly population health: a comprehensive literature review. Clin Pract Epidemiol Ment Health. 2014 Oct 21;10:103-15. doi: 10.2174/1745017901410010103. eCollection 2014. PMID 25356084
- [Result] Lara E, Olaya B, Garin N, Ayuso-Mateos JL, Miret M, Moneta V, Haro JM. Is cognitive impairment associated with suicidality? A population-based study. Eur Neuropsychopharmacol. 2015 Feb;25(2):203-13. doi: 10.1016/j.euroneuro.2014.08.010. Epub 2014 Aug 21. PMID 25190638
- [Result] Garin N, Olaya B, Lara E, Moneta MV, Miret M, Ayuso-Mateos JL, Haro JM. Visual impairment and multimorbidity in a representative sample of the Spanish population. BMC Public Health. 2014 Aug 8;14:815. doi: 10.1186/1471-2458-14-815. PMID 25103270
- [Result] Miret M, Caballero FF, Huerta-Ramirez R, Moneta MV, Olaya B, Chatterji S, Haro JM, Ayuso-Mateos JL. Factors associated with suicidal ideation and attempts in Spain for different age groups. Prevalence before and after the onset of the economic crisis. J Affect Disord. 2014 Jul;163:1-9. doi: 10.1016/j.jad.2014.03.045. Epub 2014 Apr 1. PMID 24836081
- [Result] Quintas R, Raggi A, Bucciarelli P, Franco MG, Andreotti A, Caballero FF, Olaya B, Chatterji S, Galas A, Merilainen-Porras S, Frisoni G, Russo E, Minicuci N, Power M, Leonardi M. The COURAGE Built Environment Outdoor Checklist: an objective built environment instrument to investigate the impact of the environment on health and disability. Clin Psychol Psychother. 2014 May-Jun;21(3):204-14. doi: 10.1002/cpp.1858. Epub 2013 Jul 29. PMID 23897864
- [Result] Leonardi M, Chatterji S, Koskinen S, Ayuso-Mateos JL, Haro JM, Frisoni G, Frattura L, Martinuzzi A, Tobiasz-Adamczyk B, Gmurek M, Serrano R, Finocchiaro C; COURAGE in Europe Project's Consortium. Determinants of health and disability in ageing population: the COURAGE in Europe Project (collaborative research on ageing in Europe). Clin Psychol Psychother. 2014 May-Jun;21(3):193-8. doi: 10.1002/cpp.1856. Epub 2013 Jul 24. PMID 23881690
- [Result] Perales J, Martin S, Ayuso-Mateos JL, Chatterji S, Garin N, Koskinen S, Leonardi M, Miret M, Moneta V, Olaya B, Tobiasz-Adamczyk B, Haro JM. Factors associated with active aging in Finland, Poland, and Spain. Int Psychogeriatr. 2014 Aug;26(8):1363-75. doi: 10.1017/S1041610214000520. Epub 2014 Apr 15. PMID 24735743
- [Result] Garin N, Olaya B, Perales J, Moneta MV, Miret M, Ayuso-Mateos JL, Haro JM. Multimorbidity patterns in a national representative sample of the Spanish adult population. PLoS One. 2014 Jan 20;9(1):e84794. doi: 10.1371/journal.pone.0084794. eCollection 2014. PMID 24465433
- [Result] Caballero FF, Miret M, Power M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Olaya B, Haro JM, Ayuso-Mateos JL. Validation of an instrument to evaluate quality of life in the aging population: WHOQOL-AGE. Health Qual Life Outcomes. 2013 Oct 23;11:177. doi: 10.1186/1477-7525-11-177. PMID 24152691
- [Result] Zawisza K, Galas A, Tobiasz-Adamczyk B, Chatterji S, Haro JM, Miret M, Koskinen S, Power M, Leonardi M. The validity of the instrument to evaluate social network in the ageing population: the Collaborative Research on Ageing in Europe Social Network Index. Clin Psychol Psychother. 2014 May-Jun;21(3):227-41. doi: 10.1002/cpp.1860. Epub 2013 Aug 12. PMID 23939715
- [Result] Raggi A, Quintas R, Bucciarelli P, Franco MG, Andreotti A, Miret M, Zawisza K, Olaya B, Chatterji S, Sainio P, Frisoni GB, Martinuzzi A, Minicuci N, Power M, Leonardi M. Validation of the COURAGE Built Environment Self-Reported Questionnaire. Clin Psychol Psychother. 2014 May-Jun;21(3):215-26. doi: 10.1002/cpp.1859. Epub 2013 Jul 16. PMID 23861306
- [Result] Raggi A, Quintas R, Russo E, Martinuzzi A, Costardi D, Frisoni GB, Franco MG, Andreotti A, Ojala M, Pena S, Perales J, Chatterji S, Miret M, Tobiasz-Adamczyk B, Koskinen S, Frattura L, Leonardi M. Mapping SAGE questionnaire to the International Classification of Functioning, Disability and Health (ICF). Clin Psychol Psychother. 2014 May-Jun;21(3):199-203. doi: 10.1002/cpp.1857. Epub 2013 Jul 17. PMID 23861299
- [Result] Ayuso-Mateos JL, Miret M, Caballero FF, Olaya B, Haro JM, Kowal P, Chatterji S. Multi-country evaluation of affective experience: validation of an abbreviated version of the day reconstruction method in seven countries. PLoS One. 2013 Apr 23;8(4):e61534. doi: 10.1371/journal.pone.0061534. Print 2013. PMID 23626697
- [Result] Domenech-Abella J, Lara E, Rubio-Valera M, Olaya B, Moneta MV, Rico-Uribe LA, Ayuso-Mateos JL, Mundo J, Haro JM. Loneliness and depression in the elderly: the role of social network. Soc Psychiatry Psychiatr Epidemiol. 2017 Apr;52(4):381-390. doi: 10.1007/s00127-017-1339-3. Epub 2017 Feb 2. PMID 28154893
- [Result] Olaya B, Moneta MV, Miret M, Ayuso-Mateos JL, Haro JM. Epidemiology of panic attacks, panic disorder and the moderating role of age: Results from a population-based study. J Affect Disord. 2018 Dec 1;241:627-633. doi: 10.1016/j.jad.2018.08.069. Epub 2018 Aug 16. PMID 30172214
- [Result] Olaya B, Moneta MV, Lara E, Miret M, Martin-Maria N, Moreno-Agostino D, Ayuso-Mateos JL, Abduljabbar AS, Haro JM. Fruit and Vegetable Consumption and Potential Moderators Associated with All-Cause Mortality in a Representative Sample of Spanish Older Adults. Nutrients. 2019 Aug 2;11(8):1794. doi: 10.3390/nu11081794. PMID 31382535
- [Result] Lara E, Caballero FF, Rico-Uribe LA, Olaya B, Haro JM, Ayuso-Mateos JL, Miret M. Are loneliness and social isolation associated with cognitive decline? Int J Geriatr Psychiatry. 2019 Nov;34(11):1613-1622. doi: 10.1002/gps.5174. Epub 2019 Jul 25. PMID 31304639
- [Result] Martin-Maria N, Caballero FF, Moreno-Agostino D, Olaya B, Haro JM, Ayuso-Mateos JL, Miret M. Relationship between subjective well-being and healthy lifestyle behaviours in older adults: a longitudinal study. Aging Ment Health. 2020 Apr;24(4):611-619. doi: 10.1080/13607863.2018.1548567. Epub 2018 Dec 28. PMID 30590962
- [Result] Cabello M, Borges G, Lara E, Olaya B, Martin-Maria N, Moreno-Agostino D, Miret M, Caballero FF, Haro JM, Ayuso-Mateos JL. The relationship between all-cause mortality and depression in different gender and age groups of the Spanish population. J Affect Disord. 2020 Apr 1;266:424-428. doi: 10.1016/j.jad.2020.01.162. Epub 2020 Jan 28. PMID 32056909
- [Result] Ayuso-Mateos JL, Morillo D, Haro JM, Olaya B, Lara E, Miret M. Changes in depression and suicidal ideation under severe lockdown restrictions during the first wave of the COVID-19 pandemic in Spain: a longitudinal study in the general population. Epidemiol Psychiatr Sci. 2021 Jun 2;30:e49. doi: 10.1017/S2045796021000408. PMID 34074355
- [Result] Lara E, Martin-Maria N, Miret M, Olaya B, Haro JM, Ayuso-Mateos JL. Is there a combined effect of depression and cognitive reserve on cognitive function? Findings from a population-based study. Psychol Health. 2022 Sep;37(9):1132-1147. doi: 10.1080/08870446.2021.1927030. Epub 2021 May 24. PMID 34029134
- [Result] Castelletti C, Lara E, Tobiasz-Adamczyk B, Koskinen S, Olaya B, Haro JM, Leonardi M, Kowal P, Chatterji S, Ayuso-Mateos JL, Miret M. Connecting and feeling: Associations between social factors and emotions in nine countries. Int J Psychol. 2023 Jun;58(3):282-291. doi: 10.1002/ijop.12892. Epub 2023 Feb 2. PMID 36727409
- See also: Age with health website info — http://edadconsalud.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Spanish general adult population non-institutionalized; aged 18+ years with oversampling of those aged 50+ years and those 80+ years); multi-stage stratified sampling; representative sample.
Pre-assignment Details: Respondents unable to undertake the interview because of severe cognitive or physical impairment were administered a shorter version of the questionnaire to a proxy respondent.
Groups:
- Cohort 2011: A total of 4753 persons participated at baseline between 2011 and 2012.
- Cohort 2019: 3,002 persons participated at this baseline between 2019 and 2021
Period: Overall Study
Arm/Group | Cohort 2011 | Cohort 2019
Started | 4753 | 3002
Second Wave | 2528 | 0 (Data in collection.)
Third Wave | 1577 | 0 (The third evaluation of this cohort is expected in 2025.)
Fourth Wave | 963 | 0
Completed | 963 | 0 (The new evaluation of this cohort is ongoing (july 2023) and it will be finish for the end of the year.)
Not Completed | 3790 | 3002

BASELINE CHARACTERISTICS:
Population: At the baseline, 4,753 participants were interviewed (2011 cohort), of which 2,528 were interviewed in the second wave and 1,577 in the third wave. In 2019-2021 3,002 participants were brought in (2019 cohort).
Groups:
- Cohort 2011 Sample Demographic Characteristics: The 2011 Cohort is part of a nationally representative sample of the Spanish noninstitutionalized adult population. Potential respondents were selected by a stratified, multistage, clustered area probability design, without replacement, according to the Spanish regions and population size.
- Cohort 2019 Sample Demographic Characteristics: In 2019-2021 3,002 participants were brought in (2019 cohort), using the same sample characteristics .
- Total: Total of all reporting groups
Arm/Group | Cohort 2011 Sample Demographic Characteristics | Cohort 2019 Sample Demographic Characteristics | Total
Number analyzed (Participants) | 4,753 | 3002 | 7755
Age, Categorical [Count of Participants; unit: Participants]
  number analyzed (Participants) | 4753 | 3002 | 7755
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2742 | 1,867 | 4609
  >=65 years | 2011 | 1,135 | 3146
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 4753 | 3002 | 7755
  (all) | 60.44 (16.24) | 58.19 (17.89) | 59.32 (17.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2,602 | 1,302 | 3904
  Male | 2,151 | 1,700 | 3851
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4753 | 3002 | 7755
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 4753 | 3002 | 7755
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 4753 | 3002 | 7755
Education [Count of Participants; unit: Participants]
  No education | 373 | 100 | 473
  Less than primary | 1,001 | 353 | 1354
  Primary | 1,306 | 761 | 2067
  Secondary | 562 | 428 | 990
  High School | 874 | 724 | 1598
  University+ | 572 | 460 | 1032
  Post graduate degree | 64 | 175 | 239
  missing data | 1 | 1 | 2
Marital status [Count of Participants; unit: Participants]
  Single | 680 | 495 | 1175
  Married | 2,670 | 1,666 | 4336
  Cohabiting | 175 | 127 | 302
  Separated/divorced | 346 | 306 | 652
  widowed | 882 | 408 | 1290
Health Status [Mean (Standard Deviation); unit: units on a scale] — 'Health' is the health state score between 0-100, 0 meaning the worst health and 100 the perfect health.
  units on a scale | 66.55 (13.11) | 68.95 (19.87) | 67.75 (16.49)

OUTCOME MEASURES:

1. Primary Outcome: Heath Status
Description: Measure: Health composite total score. Construct: Health status. Final result: A global total score. Range: 0-100. 0 means lower health status.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
score on a scale | 66.55 (13.11) | 68.95 (19.87)

2. Primary Outcome: Disability
Description: Measure: World Health Organization's Disability Assessment Schedule-II (WHODAS-II). Construct: Disability. Final result: A global total score. Range: 0-100. 0 means lower disability
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2011 Sample Demographic Characteristics | Cohort 2019 Sample Demographic Characteristics
Number analyzed (Participants) | 4,753 | 3,002
score on a scale | 11.17 (17.59) | 9.01 (18.20)

3. Primary Outcome: Experienced Well-being
Description: Abbreviated Version of the Day Reconstruction Method. Construct: Experienced wellbeing.
  Final Result: The used scale reports two global scores:
  * Positive Affect total score. Range: 0-100 where 0 means lower positive affect.
  * Negative Affect total score. Range 0-100 where 0 means lower negative affect.
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
score on a scale
  Positive Affect: number analyzed (Participants) | 4583 | 2911
  Positive Affect | 4.88 (1.11) | 4.75 (1.59)
  Negative Affect: number analyzed (Participants) | 4583 | 2911
  Negative Affect | 0.64 (0.89) | 0.33 (0.61)

4. Primary Outcome: Quality of Life (WHOQOL-AGE)
Description: Measure: World Health Organization Quality of Life-Age (WHOQOL-AGE) (Caballero, et al., 2013). Construct: Quality of life. Final Result: A global total score. Range 0-100. 0 means lower quality of life
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4583 | 2,892
score on a scale | 72.30 (14.90) | 76.17 (15.25)

5. Secondary Outcome: Number of Participants With Depression
Description: Measure: The World Health Organization Composite International Diagnostic Interview (CIDI). Depression module (WHO-CIDI, 1990).
  Construct: Presence of Depression. Final result: Two measures of depression according to Research Diagnostic Criteria.
  * Presence of 12 month depression. Values (yes/no).
  * Presence of lifetime depression. Values (yes/no).
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4583 | 2911
Participants | 510 | 203

6. Secondary Outcome: Presence of Suicide Behavior
Description: Measure: The World Health Organization Composite International Diagnostic Interview (CIDI). Suicide module (WHO-CIDI, 1990).
  Construct: Presence of Suicide behavior The instrument reports six measures of suicide behavior.
  * Presence of 12 month suicide ideation. Values (yes/no)
  * Presence of 12 month suicide planning. Values (yes/no)
  * Presence of 12 month suicide attempts. Values (yes/no)
  * Presence of lifetime suicide ideation. Values (yes/no)
  * Presence of lifetime suicide planning. Values (yes/no)
  * Presence of lifetime suicide attempts. Values (yes/no)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
Participants | 161 | 75

7. Secondary Outcome: Presence of Anxiety Disorders
Description: Measure: The World Health Organization Composite International Diagnostic Interview (CIDI). Anxiety disorders module (WHO-CIDI, 1990).
  Construct: Presence of anxiety Disorders Final Result: The instrument included in the study reports six measures of anxiety disorders according to Research diagnostic criteria.
  * Presence of 12 month panic disorder. Values (yes/no)
  * Presence of 12 month generalized anxiety disorder. Values (yes/no)
  * Presence of 12 month phobic disorder. Values (yes/no)
  * Presence of lifetime panic disorder. Values (yes/no)
  * Presence of lifetime generalized anxiety disorder. Values (yes/no)
  * Presence of lifetime phobic disorder. Values (yes/no)
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4583 | 3,002
Participants | 69 | 77

8. Secondary Outcome: Presence of Diabetes
Description: Construct: Presence of diabetes Measure: Self-reported information of 12-month presence of diagnosis and/or of treatment for diabetes Values: (Yes/No)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4,753 | 3,002
Participants | 661 | 353

9. Secondary Outcome: Presence of Lung Disease
Description: Construct: Presence of any lung disease Measure: Self-reported information of 12-month presence of diagnosis and/or of treatment for any lung disease Values: (Yes/No)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
Participants | 399 | 152

10. Secondary Outcome: Presence of Stroke
Description: Construct: Presence of stroke Measure: Self-reported information of 12-month presence of diagnosis and/or of treatment for stroke Values: (Yes/No)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
Participants | 183 | 82

11. Other Pre Specified Outcome: Alcohol Use Information
Description: Construct: Alcohol use Measure: Self-reported information of how many standard drinks per day in last 7 days have been used.
  Values: four categories of alcohol use:
  0= Lifetime abstainers: Participants that have never used alcohol
  1. Occasional drinkers: Participants that have ever used alcohol but not in the previous 7 days
  2. Non-heavy drinker: Participants did consume alcohol in the last 30 days and in the last 7 days
  3. Infrequent heavy drinker: Participants did consume alcohol 1-2 days per week, with 5 or more standard drinks per day in last 7 days for men and 4 or more standard drinks per day in last 7 days for women.
  4. Frequent heavy drinkers: Participants did consume alcohol 3 or more days per week with 5 or more standard drinks per day in last 7 days for men and 4 or more standard drinks per day in last 7 days for women.
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4583 | 2911
Participants
  Lifetime abstainers | 1,345 | 871
  Occasional drinkers | 1,424 | 1,055
  Non-heavy drinker | 1,671 | 846
  Infrequent heavy drinker | 111 | 95
  Frequent heavy drinker | 32 | 38
  Missing | 0 | 6

12. Other Pre Specified Outcome: Tobacco Use Information
Description: Construct: Tobacco use Measure: Self-reported information of how many cigarettes/pipes/tobacco products/ have been used in the last week.
  Values: Four categories of tobacco use:
  0= Never smokers: Participants who have never used tobacco
  1. Daily smokers: Participants who have used tobacco last week
  2. Non daily smokers: Participants who have ever used tobacco but not in the previous week
  3. Former smokers: Participants who smoked in the past (ex smokers)
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4583 | 2911
Participants
  Never smokers | 2,339 | 1,543
  Daily smokers | 1,049 | 626
  Non daily smokers | 100 | 52
  Former smokers | 1095 | 690

13. Other Pre Specified Outcome: Level of Physical Activity
Description: Construct: Level of physical activity Scale: Global Physical Activity Questionnaire version 2 (GPAQ v2); It collects information on physical activity participation in three settings (or domains) and sedentary behavior. The responses given by the participants have been converted to Metabolic Equivalent to Task (MET) values. Applying MET values to activity levels allows for calculating total physical activities.
  Values: Three values of physical activity can be obtained 3=High physical activity 2=Moderate physical activity
  1=Low physical activity
Time Frame: Baseline
Population: Proxy respondent were not analysed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4583 | 2902
Participants
  high | 1,464 | 898
  Moderate | 1,724 | 1,013
  Low | 1,395 | 991

14. Other Pre Specified Outcome: Level of Social Support
Description: Construct: Social Support Measure: 3-Item Oslo Social Support Scale (OSLO) (Abiola et al., 2013) Result: A global total score, then transformed into a percentile scale. Range: 0-100. Higher scores indicate a higher social support.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
score on a scale | 77.50 (16.73) | 77.44 (17.70)

15. Other Pre Specified Outcome: Intensity of Subjective Perception of Loneliness
Description: Construct: Loneliness Measure: Three-item University of California, Los Angeles (UCLA) Loneliness Scale (Hughes et al, 2004) Result: A total loneliness score, then transformed into a percentile scale. Range: 0-100. Higher scores means higher loneliness
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2011 | Cohort 2019
Number analyzed (Participants) | 4753 | 3,002
score on a scale | 12.34 (24.25) | 10.74 (22.82)

ADVERSE EVENTS:
Time Frame: For both cohorts (2011 and 2019), data on adverse events and deaths are collected at the same time, when a new wave is carried out. Specifically for cohort 2011 adverse events have been evaluated 4 times during 12 years (2011-2012, 2014-2015, 2019-2021 and 2022-2023) and for cohort 2019 they have been evaluated 2 times during 4 years (2019-2020 and 2022-2023).
Description: Diverse chronic conditions were assessed through self-reported physician's diagnosis, symptom-based algorithms (e.g., stroke, chronic obstructive lung disease - COPD), and/or measurements to detect undiagnosed cases. This section also included questions on treatments and age of onset
Groups:
- Cohort 2011: The data comprising the 2011 reference cohort were collected as part of the Collaborative Research on Ageing in Europe (COURAGE in Europe) project between July 2011 and May 2012. It consisted of a representative sample of the Spanish adult population over 50 years of age, with an oversampling of older people and a representative comparison sample of individuals aged 18-49 years. Potential respondents were selected using a stratified, multistage, stratified probability design, by clustered areas without replacement, according to Spanish regions and population size. The primary sampling unit consisted of municipalities. A number of census units (the secondary sampling unit) were chosen from each of them. Age strata were then used to randomly select 10 households within each census unit (the tertiary sampling unit). Finally, a list of household occupants was drawn up, from which one participant was randomly selected following age quotas. Institutionalized persons were not included in the initial interviews. At baseline, 4,753 participants were interviewed, of which 2,528 were interviewed in the second wave (2014-2015), 1,577 in the third wave (2010-2021) and 963 in the fourth wave (2022-2023).
- Cohort 2019: The sample of the 2019 cohort is a new representative refreshment sample from the provinces of Barcelona and Madrid, to compensate for attrition (e.g., deaths, dropouts) from the 2011 cohort. Household selection was also multistage. At the primary sampling unit level, households were defined using predefined routes and an omission factor. Households were assigned to one of two age groups (i.e., household aged 18-49 years or household aged 50 years or older) and interviewers hand-delivered the invitation letter to the selected households. All residents in the eligible age group were invited to participate in the survey. In this first wave, 3 002 participants joined and in 2022 the second selection of participants for the 2019 cohort was conducted, of which 1 037 participants were interviewed.
Arm/Group | Cohort 2011 | Cohort 2019
All-Cause Mortality (participants affected / at risk) | 591/4753 | 157/3002
Serious Adverse Events (participants affected / at risk) | 706/4753 | 234/3002
Other Adverse Events (participants affected / at risk) | 1447/4753 | 1474/3002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 2011 (N=4753) | Cohort 2019 (N=3002)
Stroke (Vascular disorders) | 280 | 82 — Participants were asked if they have had a stroke diagnosed by a doctor. Other related questions were asked, as if the participants suffered from sudden paralysis of legs or arms of one side of his body.
Lungs problems (Respiratory, thoracic and mediastinal disorders) | 426 | 152 — Participants were asked if they ever have been diagnosed of some chronic lungs illness, as emphysema, chronic bronchitis, chronic obstructive lungs illness), and related questions, as if they feel lack of breathing in the last 12 months.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 2011 (N=4753) | Cohort 2019 (N=3002)
Arthritis (Musculoskeletal and connective tissue disorders) | 808 | 794
Diabetes (Metabolism and nutrition disorders) | 325 | 353
Cataract (Eye disorders) | 314 | 327 — Vision Problem

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No